CLINICAL TRIAL: NCT04217109
Title: KDOG1 :Transcutaneous Breast Cancer Diagnosis by Canine Odorology
Brief Title: Transcutaneous Breast Cancer Diagnosis by Canine Odorology
Acronym: KDOG1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A01592-55
Record Dates: First submitted 2019-11-19; First posted 2020-01-03 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Dog Detection; Volatile organic Compounds
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Odour sampling (Experimental): Odour collection will be obtained by positioning a compress on the breast concerned during the night preceding the day of samplings. The compress, once removed, will be placed in specific envelope for the study. Envelope will be given to the investigating centre during the appointment of percutaneous samples and then sent to the sponsor center (Institute Curie Paris).
  Interventions: Diagnostic Test: Odour sampling

INTERVENTIONS:
Diagnostic Test: Odour sampling — Upon receipt of the samples at the Institute Curie-Paris, the compresses will be packed in jars and then transmitted to the dog center and analyzed by the study dogs.
  Positive marking is characterized by a sitting position of the dog in front of the sample.

SUMMARY:
Patient with an indication of interventional percutaneous procedure for characterization of a breast lesion, palpable or not, classified as category 4 or 5, according to the Breast Imaging (BI) Report and Data System of the American College of Radiology (RADS) classification detected at mammography and/or breast ultrasound examination.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years and older, with one or more ipsilateral mammary lesion(s), palpable or not, detected at mammography and/or ultrasound and with at least one lesion classified as BI-RADS® category 4 or 5 with an indication of percutaneous sampling (cytology, microbiopsies, macro-biopsies) ;
2. Benefit from the national social security ;
3. Signature of the informed consent of the study ;
4. There is no contraindication for the person to simultaneously participate to another research program and there is no exclusion period planned after the study.

Exclusion Criteria:

1. Patient with bilateral breast lesions classified as BI-RADS® category 4 or 5;
2. Patient with breast implant(s);
3. Patient with a personal history of breast surgery for benign lesion(s) of the concerned breast operated less than 4 weeks before the date of inclusion in this study;
4. Patient with a personal history of cancer (in situ or invasive) less than 5 years before inclusion whatever the anatomical site including cutaneous basal cell carcinoma;
5. Patient with a personal history of punctures and/or percutaneous breast biopsies of the concerned breast less than 4 weeks before inclusion;
6. Patient with a breast skin ulceration;
7. Patient under insulin (risk of sudation that may impair compress sample);
8. Concomitant antibiotics or corticoids taken one week before inclusion in the study;
9. Patient with a current viral infection (fever);
10. Persons under guardianship or deprived of liberty;
11. Impossibility to submit to the medical monitoring expected by the study for geographical or severe psychological reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Evaluate the sensitivity and specificity of canine odorology in women with breast lesion | 26 months
  The sensitivity and specificity of canine odorology in women with undeterminate breast lesion classified American College of Radiology (ACR) 4 or 5 (typically malignant) will be compared to the anatomopathological results of breast percutaneous sampling (biopsy)

SECONDARY OUTCOMES:
Sensitivity (markings on patients affected) and specificity (no-markings on patients not affected) | 38 months
  Number of markings among compresses of patients affected and number of no-markings among compresses of patients not affected. The gold standard is the pathological examination of the operative specimen or the status of the patient at 1 year.
Positive predictive value (PPV) and negative predictive value (NPV) of canine odorology | 38 months
  Number of compresses of patient affected on number of markings (PPV) and number of compresses of patient non affected on number of no-markings (NPV) will be evaluated
Patient compliance during the study | 26 months
  The rate of return of compresses after delivery of a kit will be evaluated
Comparison between canine odorology and mammography | 38 months
  Comparison test of sensitivity and specificity values between canine odorology and mammography
Performance of each dog | 26 months
  Sensitivity and specificity of canine odorology for each dog will be calculated
Variability between dogs | 26 months
  A Cohen's kappa test will be used to explore the variability between trained dogs and dog breeds
Performance of canine odorology if the test is based on 2 dogs | 24 months
  The results of the 2 dogs will be used to compare the performances
Patient's satisfaction | 26 months
  A questionnaire will be completed by the patients to measure their satisfaction and indicate their level of agreement. A score from 0 (no anxiety) to 5 (very anxious) on a scale will be completed to assess anxiety, a score from 0 (very difficult) to 5 (very easy) will be used to ensure that the compress is easy to use.

CONTACTS AND LOCATIONS:
Overall Officials: ANNE TARDIVON, MD, Principal Investigator — Institut Curie
Locations (7):
- France (7):
  - Centre République, Clermont-Ferrand
  - Centre Hospitalier Universitaire, Limoges
  - Institut de Cancérologie de l'Ouest, Nantes
  - Groupe Hospitalier Paris Saint- Joseph, Paris
  - Institut Curie, Paris
  - Institut Curie, Saint-Cloud
  - Centre Hospitalier Valenciennes, Valenciennes